CLINICAL TRIAL: NCT03488368
Title: Quality Control of STOP-IgAN Trial Results in Longterm Observation With Existing Routine Data of Randomized Trial Participants (STOP-IgAN - Longterm) - Observational Study
Brief Title: Longterm Renal Oucomes of STOP-IgAN Trial Participants
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jürgen Floege, Prof. Dr. Jürgen Floege, RWTH Aachen University
Other Study IDs: STOP IgAN - Longterm
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Supportive-care group: Observation of IgAN patients who received supportive care measures (without additional immunosuppression) during the first three years after randomization, i.e. trial phase of the original STOP-IgAN trial.
  Interventions: Other: observation
- Immunosuppression group: Observation of IgAN patients who received supportive care measures and additional immunosuppression during the first three years after randomization, i.e. trial phase of the original STOP-IgAN trial.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Observation of renal outcome parameters and adverse events in the follow-up beyond the 3-year trial phase of the original STOP-IgAN trial.

SUMMARY:
IgA nephropathy (IgAN) is the most prevalent form of primary glomerulonephritis in the Western world. Although most IgAN patients take a benign longterm course, about 20-30% progress to end-stage renal disease (ESRD) over 20 years. The majority of current treatment recommendations is based on weak evidence.

In the randomized, controlled Supportive Versus Immunosuppressive Therapy for the Treatment Of Progressive IgAN (STOP-IgAN) trial, the investigators analyzed whether additional immunosuppression on top of standardized supportive care provides renal benefits in patients with progressive IgAN. Patients with persisting proteinuria >0.75 g/d (n=162) despite optimized supportive treatment including control of blood pressure and proteinuria, were randomized to either continue on supportive care or to receive additional immunosuppression during the 3-year trial phase. It was observed that immunosuppressive therapy in addition to optimized supportive care led to more full clinical remissions, but eventually did not better preserve renal function, did not better save patients from ESRD development and evoked more adverse effects such as infections, weight gain and diabetes.

Aim of this planned study is to analyze renal outcome measures and adverse effects in the longterm observation of all randomized STOP-IgAN participants to ascertain quality and strength of the original trial results. By its observational nature, this quality control study includes the 162 IgAN patients (with the exception of drop-out patients) that had been previously randomized into the original STOP-IgAN trial.

Information on serum creatinine, proteinuria, ESRD, death, relevant adverse events such as major cardiovascular events, osteoporosis, osteonecrosis, bone fractures, diabetes, malignancies and interim treatment will be collected as available from existing routine records until March 31, 2018.

Primary endpoint is the time to the first occurring event of the binary composite of all-cause death, ESRD or decline in estimated glomerular filtration rate (eGFR) by at least 40% as compared to enrollment into the original trial. Secondary outcome measures comprise the individual components of the primary endpoint, absolute eGFR at the end of observation, proteinuria and adverse events. Information on specific treatments with renin-angiotensin-system (RAS)-blocking agents and/or interim immunosuppression will also be collected. All data will be recorded in a pseudonymous fashion in a central electronic data base located at the PI's site.

DETAILED DESCRIPTION:
Aim: Observational quality control study to analyze renal outcome measures and adverse events in the longterm observation of all randomized STOP-IgAN participants to ascertain quality and strength of the original trial results.

Eligible subjects/sample size: By its observational nature, this study includes the 162 IgAN patients (with the exception of drop-out patients) that had been previously randomized into the original STOP-IgAN trial. Since this study is performed as quality control study of previously randomized patients, a new written informed consent is not necessary.

Endpoints: Primary endpoint is the time to the first occurring event of the binary composite of all-cause death, ESRD or decline in estimated glomerular filtration rate (eGFR) by at least 40% as compared to enrollment into the original trial (time-to-event analysis). Secondary outcome measures comprise the individual components of the primary endpoint, absolute eGFR at the end of observation, proteinuria and adverse events. Information on specific treatments with renin-angiotensin-system (RAS)-blocking agents and/or interim immunosuppression will also be collected.

Data collection: Available information on serum creatinine, proteinuria, ESRD, death, relevant adverse events such as major cardiovascular events, osteoporosis, osteonecrosis, bone fractures, diabetes, malignancies and interim treatment will be collected retrospectively as available from existing nephrology routine records until March 31, 2018. The involved nephrology departments (all in Germany) will be contacted by phone and asked to provide these informations from the randomized STOP-IgAN patients. All data will be recorded in a pseudonymous fashion in a central electronic data base located at the PI's site. To assure high-standard data quality, source data entry will be performed in a double-entry mode, i.e. each data point will be entered independently by two individuals.

ELIGIBILITY:
Inclusion Criteria:

All randomized STOP-IgAN participants.

Exclusion Criteria:

Drop-outs of the main STOP-IgAN trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All randomized STOP-IgAN participants with the exception of drop-outs.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Time to the first occurring event of the binary composite of all-cause death, end-stage renal disease (ESRD) and of estimated glomerular filtration rate (eGFR)-loss >40% based on available data by March 31, 2018. | as available by March 31, 2018
  Time to the first occurring event of the binary composite of all-cause death, end-stage renal disease (ESRD) and of estimated glomerular filtration rate (eGFR)-loss >40% based on available data by March 31, 2018. For GFR-loss, we consider eGFR values baseline (enrolment into original STOP-IgAN trial) and the last two available values by March 31, 2018. For GFR-loss, eGFR will be calculated using the creatinine-based, formula of Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi). Data will be considered at baseline, 6 months, 12 months, 24 months and 36 months after randomization and the last two available values by March 31, 2018.

SECONDARY OUTCOMES:
all-cause death | as available by March 31, 2018
  death by any cause.
end-stage renal disease (ESRD) | as available by March 31, 2018
  date of first occurrence of ESRD, i.e. initiation of regular dialysis therapy or renal transplant
first occurrence of eGFR-loss > 40% | as available by March 31, 2018
  Values will be considered of the first three years after randomization and the last two available values by March 31, 2018.
first occurrence of eGFR-loss > 30% | as available by March 31, 2018
  Values will be considered of the first three years after randomization and the last two available values by March 31, 2018.
course of proteinuria | as available by March 31, 2018
  Values will be considered of the first three years after randomization and the last two available values by March 31, 2018.
Occurrence of major adverse cardiovascular events (MACE) and other relevant adverse events | as available by March 31, 2018
  MACE included one of the following events: cardiovascular death, myocardial infarction, transient ischemic attack (TIA), stroke, peripheral vascular event.
  Other relevant side effects include diabetes mellitus, osteoporosis, osteonecrosis, bone fracture, malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Floege, MD, Principal Investigator — RWTH Aachen University, University Hospital
Locations (1):
- Medical Clinic II, University Hospital Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rauen T, Eitner F, Fitzner C, Sommerer C, Zeier M, Otte B, Panzer U, Peters H, Benck U, Mertens PR, Kuhlmann U, Witzke O, Gross O, Vielhauer V, Mann JF, Hilgers RD, Floege J; STOP-IgAN Investigators. Intensive Supportive Care plus Immunosuppression in IgA Nephropathy. N Engl J Med. 2015 Dec 3;373(23):2225-36. doi: 10.1056/NEJMoa1415463. PMID 26630142